CLINICAL TRIAL: NCT07271134
Title: Short-term Observation on the Clinical Application Effect of Astra Tech Implant EV Short Implants for Maxillary Sinus Elevation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linhu Wang (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor-Investigator, Linhu Wang, Medical professor, Wuhan Central Hospital
Organization: Wuhan Central Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WHZXKYL2025-123; I-AS-25-105 (Other Grant/Funding Number: DENTSPLY IH AB)
Record Dates: First submitted 2025-11-22; First posted 2025-12-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Missing Teeth
Keywords: Short implant; Maxillary sinus floor elevation
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- transcrestal sinus floor elevation (Experimental)
  Interventions: Device: short implants (L=6.3mm); Procedure: short implants (L=8mm); Device: conventional implants (L=9mm)

INTERVENTIONS:
Device: short implants (L=6.3mm) — Short-term clinical outcome of Astra OsseoSpeed EV short implants (L=6.3mm) for transcrestal sinus floor elevation
Procedure: short implants (L=8mm) — Short-term clinical outcome of Astra OsseoSpeed EV short implants (L=8mm) for transcrestal sinus floor elevation
Device: conventional implants (L=9mm) — conventional implants (L=9mm) in the posterior maxillary region for dental restoration

SUMMARY:
Short-term comparison of clinical application effects of Astra OsseoSpeed EV short implants and conventional implants for maxillary sinus elevation

DETAILED DESCRIPTION:
1. If the survival rate, marginal bone resorption , complications and patient satisfaction of the short implant group are comparable or better than those of the conventional implant group, then short implants can be regarded as an effective treatment option for insufficient alveolar bone in the posterior teeth area. Thus, in clinical practice, the investigators can utilize short implants combined with transcrestal sinus floor elevation, or even implant short implants to help patients with certain insufficient maxillary bone complete implant restoration without resorting to more complex, costly and more invasive external elevation surgery to increase the length of posterior teeth implants in the maxillary region.
2. If it is found that the short implant group has a higher incidence of complications or a lower long-term survival rate, further exploration of its indications and optimization of surgical strategies is required.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old with at least one area of the posterior dental arch having insufficient alveolar bone height (3-6 mm)
* Patients are in good health and have no major systemic diseases such as diabetes or cardiovascular diseases, and no maxillary sinus lesions
* They are willing to undergo implant restoration treatment and can complete at least 3-year follow-up.

Exclusion Criteria:

* horizontal bone deficiency alveolar ridges,bone defects caused by tumor resection
* excessive tobacco use (more than 10 cigarettes per day)
* severe liver and kidney diseases
* history of radiotherapy and chemotherapy in the head and neck region
* uncontrolled diabetes
* active periodontal disease
* oral mucosal diseases in the treatment area or poor oral hygiene,
* PI > 70%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Various complications | From having a tooth implant to one year after wearing the dentures
  the rate of Implant survival, swelling, pain, etc.

SECONDARY OUTCOMES:
marginal bone resorption | one year
  Measure the changes in the bone height around the implant

OTHER OUTCOMES:
Patient satisfaction | From having a tooth implant to one year after wearing the dentures
  Very satisfied, satisfied, dissatisfied, the rate of dissatisfaction, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 26, Shengli Street, Jiang'an District, Wuhan City, Hubei Province, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Methods and Results
Supporting Information: Study Protocol, ICF, CSR